CLINICAL TRIAL: NCT00000420
Title: Safety of Estrogens in Lupus Erythematosus - National Assessment (SELENA): Oral Contraceptives
Brief Title: Safety of Estrogens in Lupus: Birth Control Pills
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Office of Research on Women's Health (ORWH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: U01 AR42540 NIAMS-028B; U01AR042540 (NIH)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; SELENA; Oral contraceptives; The pill; Birth control; Condom; Diaphragm; Estrogen; Lupus; Placebo
MeSH Terms: conditions — Lupus Erythematosus, Systemic

INTERVENTIONS:
Drug: Ortho-Novum 777

SUMMARY:
Safety of Estrogens in Lupus Erythematosus - National Assessment (SELENA) is a study to test whether women with systemic lupus erythematosus (SLE or lupus) can safely use estrogen. We will determine this by looking at the effects of oral contraceptives (birth control pills, also known as "the pill") on disease activity and severity in women with SLE. The results of the study will show whether it is safe for women with SLE to use the pill.

DETAILED DESCRIPTION:
This study tests the effect of exogenous female hormones on disease activity and severity in women with systemic lupus erythematosus (SLE). Physicians generally do not prescribe oral contraceptives (OCs) to women with lupus because of the widely held view that these drugs can activate SLE. This practice is based on the greater incidence of SLE in women than in men, biologic abnormalities of estrogen metabolism, murine models of lupus, several anecdotes of patients having disease flares while receiving exogenous hormones, and a single retrospective study in patients with preexisting renal disease.

By contrast, recent retrospective studies suggest that the rate of flare is not significantly increased in patients taking OCs. The preexisting data is insufficient to warrant the dismissal of a potentially important birth control option in a disease that predominantly affects women in their reproductive years and whose fertility is not altered by the disease. Moreover, the use of OCs to preserve fertility in patients taking cyclophosphamide and the use of estrogens to prevent coronary artery disease and postmenopausal and steroid-induced osteoporosis are timely considerations.

We will attempt to define, in a multicenter, randomized, double-blind, placebo-controlled trial, the effect of OCs containing low-dose synthetic estrogens and progestins on disease activity in women with SLE. Because the research hypothesis is that OCs do not increase the risk of flares, we have designed the study to be able to detect minimal increases in the rate of flares in patients taking OCs.

We will enroll patients with inactive, stable, or moderate disease requiring less than 0.5 mg prednisone per kg of bodyweight per day over a 2-year period and randomize them to receive birth control pills or placebo pills for 12 months. During that time, the patient must use condoms or a diaphragm as birth control. We will recruit patients from clinics and private practices that include over 4,000 women with SLE, most belonging to minority groups.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Unequivocal diagnosis of SLE
* Inactive disease or be stable on 0.5 mg/kg/day or less of predisone
* Must be between 18 and 39 years old if non-smoker
* Must be between 18 and 35 years old if smoker

Exclusion Criteria:

* Blood pressure >145/95 on three occasions
* Deep vein, arterial thrombosis or pulmonary embolus
* GPL >40; MPL >40; APL >50; dRVVT >37 sec
* APL antibody syndrome ever
* Gynecologic or breast cancer
* Hepatic dysfunction or liver tumors
* Diabetes mellitus (NOT due to steroids) with vascular disease
* Congenital hyperlipidemia
* Complicated migraine
* Severe disease activity (SLEDAI >12)
* Increase in SLEDAI >2 points in 3 months
* Unexplained vaginal bleeding
* Use of estrogen (OCP) for >1 month at any time after SLE diagnosis
* Present pregnancy
* Angina or MI due to APS
* Age >35 yrs. for smokers; >39 yrs. for nonsmokers

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350
Dates: Start 1997-06; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Jill P. Buyon, MD, Principal Investigator — Hospital for Joint Diseases; Michelle Petri, MD, Study Director — Johns Hopkins University Hospital, Dept. of Rheumatology
Locations (15):
- United States (15):
  - UCLA Medical Center, Dept. of Rheumatology, Los Angeles, California
  - University of Chicago Pritzker School of Medicine, Chicago, Illinois
  - Louisiana School of Medicine, Dept. of Medicine/Immunology, Shreveport, Louisiana
  - Johns Hopkins Hospital, Dept. of Rheumatology, Baltimore, Maryland
  - Univ. of Michigan Med. Ctr., Rheumatology Division, Ann Arbor, Michigan
  - Hospital for Joint Diseases, New York, New York
  - Hospital for Special Surgery, Dept. of Rheumatology, New York, New York
  - Albert Einstein College of Medicine, Jacobi Hospital, Dept. of Rheumatology, The Bronx, New York
  - UNC Medical Center, Dept. of Rheumatology, Chapel Hill, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Univ. of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Univ. of Pittsburgh, Dept. of Rheumatology, Pittsburgh, Pennsylvania
  - University of Texas Health Sciences Center, Houston, Texas
  - Medical College of Virginia, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Buyon JP. Clinical trials in systemic lupus erythematosus. Curr Rheumatol Rep. 2000 Feb;2(1):11-12. doi: 10.1007/s11926-996-0062-y. No abstract available. PMID 11123033
- [Background] Petri M, Buyon J, Kim M. Classification and definition of major flares in SLE clinical trials. Lupus. 1999;8(8):685-91. doi: 10.1191/096120399680411281. PMID 10568907
- [Background] Kim MY, Buyon JP, Petri M, Skovron ML, Shore RE. Equivalence trials in SLE research: issues to consider. Lupus. 1999;8(8):620-6. doi: 10.1191/096120399680411308. PMID 10568898
- [Background] Buyon JP, Dooley MA, Meyer WR, Petri M, Licciardi F. Recommendations for exogenous estrogen to prevent glucocorticoid-induced osteoporosis in premenopausal women with oligo- or amenorrhea: comment on the American College of Rheumatology recommendations for the prevention and treatment of glucocorticoid-induced osteoporosis. Arthritis Rheum. 1997 Aug;40(8):1548-9. doi: 10.1002/art.1780400831. No abstract available. PMID 9259444
- [Background] Buyon JP. Oral contraceptives in women with systemic lupus erythematosus. Ann Med Interne (Paris). 1996;147(4):259-64. PMID 8952745
- [Background] Buyon JP, Wallace DJ. The endocrine system, use of exogenous estrogens, and the urogenital tract. In Dubois' Lupus Erythematosus, 6th edition. Wallace DJ, Hahn BH, eds. Philadelphia: Lippincott Williams & Wilkins, 2002; pp. 821-841.
- [Background] Buyon JP. Hormone replacement therapy in postmenopausal women with systemic lupus erythematosus. J Am Med Womens Assoc (1972). 1998 Winter;53(1):13-7. PMID 9458619
- [Result] Petri M, Kim MY, Kalunian KC, Grossman J, Hahn BH, Sammaritano LR, Lockshin M, Merrill JT, Belmont HM, Askanase AD, McCune WJ, Hearth-Holmes M, Dooley MA, Von Feldt J, Friedman A, Tan M, Davis J, Cronin M, Diamond B, Mackay M, Sigler L, Fillius M, Rupel A, Licciardi F, Buyon JP; OC-SELENA Trial. Combined oral contraceptives in women with systemic lupus erythematosus. N Engl J Med. 2005 Dec 15;353(24):2550-8. doi: 10.1056/NEJMoa051135. PMID 16354891